CLINICAL TRIAL: NCT00344487
Title: The Effect of Kaletra on CD4 Immune Reconstitution in HIV-infected Patients With Long-term Virologic Suppression on a Non-Kaletra Containing ART Regimen, But With a Blunted Immune Response
Brief Title: Pilot Study of Effect of Kaletra on CD4 Response in HIV Positive (+) Patients With Viral Suppression KIMBO Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to enroll subjects.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Mohammad Sajadi, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-27050
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: HIV
MeSH Terms: interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lopinavir/ritonavir (Kaletra) (Experimental): lopinavir/ritonavir (Kaletra)400/100mg tablets by mouth twice a day for 48 weeks.
  Interventions: Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Lopinavir/Ritonavir — Dosing of Kaletra will be per package insert and BID with food. A three-drug standard of care antiretroviral regimen will be used in this study. Subjects will enter the study already on an effective, virally-suppressive treatment regimen. One of these drugs will be substituted for Lopinavir/ritonavir (Kaletra®). However, the nucleoside/nucleotide backbone drugs that the subject is already on will remain the same.
  Other Names: Kaletra

SUMMARY:
To explore the hypothesis that the use of Lopinavir/ritonavir will be associated with improved CD4 immune reconstitution in volunteers who fail to demonstrate a significant CD4 cell increase (while on their first antiretroviral treatment regimen) despite sustained viral suppression by a non-Lopinavir/ritonavir-containing regimen

DETAILED DESCRIPTION:
This is an open-labeled, non-randomized exploratory trial in selected volunteers who meet the stated enrollment criteria. This study will assess the impact of Lopinavir/ritonavir on CD4 immune reconstitution. All volunteers must have been on antiretroviral therapy with sustained viral load suppression of < 400 copies/mL for at least 24 months (or, HIV-1 RNA < 400 copies/mL for 12 months, during which HIV-1 RNA was < 50 copies/mL for 6 months prior to screen). Despite induction of viral suppression, all volunteers must have demonstrated limited post-antiretroviral CD4 increase.

Lopinavir/ritonavir will be substituted for one of the 3 ARV drugs in the current (baseline) antiretroviral treatment regimen. Lopinavir/ritonavir will be substituted for any of the following: 3rd NRTI, an NNRTI, a PI or a boosted PI, while the nucleoside backbone will remain the same. If the subject is currently on a three-drug nucleoside/nucleotide plus a 4th anchor drug such as a NRTI, NNRTI, PI or boosted PI regimen, the triple nucleoside will remain constant and only the anchor drug is to be substituted with Lopinavir/ritonavir. Patients on 2 NRTIs with an NNRTI and a PI combination will not be allowed in the study.

Patients will be evaluated frequently, to include physical examination, assessment for the development of AIDS-defining conditions, hematology, chemistry, lipid profile, CD4 CD8 cell counts, plasma HIV-1 RNA ultrasensitive, and assessment of adverse events. If HIV-1 RNA becomes detectable, this will be repeated for confirmation with 2 weeks. HIV genotyping and phenotyping will be performed on patients who demonstrate repetitive plasma viral load levels of > 1,000 copies/mL.

An assessment of memory and naïve T cell response to antiretroviral regimen change will be performed in this study.

Dose and dose selection Lopinavir/ritonavir is also approved for once a day dosing. The dose of lopinavir/ritonavir (Kaletra) for this study will be 400/100mg. BID or 800/200mg. qd. New tablet formulation no longer requires that lopinavir/ritonavir be taken with food. We will give the volunteer the option for once a day dosing or BID dosing of Kaletra. However, those switching from an NNRTI to Kaletra will initially be placed on BID dosing of Kaletra, and allowed to switch to once-a-day dosing of Kaletra after 4 weeks on study drug.

ELIGIBILITY:
Inclusion criteria

1. Human Immunodeficiency Virus type-1 (HIV-1)infection, as documented by any licensed enzyme-linked immunosorbent assay ELISA)test kit, and confirmed by Western blot, positive HIV-1 blood culture, positive HIV serum antigen, or plasma viremia at any time prior to study entry. If no record exists, testing must occur at screening.
2. Males and non-pregnant females > 18 years of age.
3. Currently on a stable antiretroviral regimen for at least 6 months prior to enrollment. This stable regimen must be their first treatment regimen, however, prior changes could have been made for toxicity or intolerability, or where providers were using an "induction /maintenance"type of treatment strategy.
4. HIV-1 RNA < 400 copies/ml (or <500 copies/ml for the bDNA test or <40 copies/ml for the nucleic acid sequence based amplification [NASBA test]) for at least 24 months; and an HIV-1 RNA < 50 copies/ml at screening; interim, non-consecutive viral load blips of < 1,000 copies/mL will be allowed
5. Or, HIV-1 RNA < 400 copies/ml (or <500 copies/ml for the bDNA test or <40 copies/ml for the NASBA test)for minimum of 12 months, during which the HIV-1 RNA was < 50 copies/ml (or <500 copies/ml for the bDNA test or <40 copies/ml for the NASBA test) for 6 months prior to screening, and < 50 copies/mL at screen
6. At a minimum of twelve months post-initiation of antiretroviral therapy, CD4 count remains < 200 cells/mm3, or if baseline CD4 count was between 200-300, and there is an increase of < 50 cells/mm3 over a 12 month period.
7. Laboratory tests within pre-specified limits
8. Able to sign the informed consent, and is willing to comply with the requirements of this clinical trial.
9. Available for at least 48 weeks of follow up.
10. If female and of child bearing potential must consent to using at least two forms of contraception
11. Participant must have a Primary Care Provider in order to be enrolled in this study.

Exclusion criteria

1. Pregnant or breast-feeding woman
2. Current treatment for malignancy other than basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or isolated cutaneous Kaposi's Sarcoma that is not being treated; those with prior cancer diagnosis, such as lymphomas must have been disease-free for at least 5 years
3. Absolute neutrophil count < 500, platelet count < 50,000, hemoglobin < 8 gm/dL
4. Evidence of end-organ disease, defined as follows: renal (calculated creatinine clearance of less than 50 mL/min); liver (liver-associated enzymes > 3 times the upper limits of normal)
5. Grade 3 (ACTG Grading Scale) or higher cholesterol or triglyceride elevations
6. Acute, serious infection requiring prescription drug therapy within 30 days prior to study entry
7. In the opinion of the investigator, there is evidence of an active ongoing opportunistic infection
8. Must not currently be undergoing treatment for an opportunistic infection.
9. Use of immune stimulation agents known to impact CD4 cell count in the peripheral circulation, to include Interleukin 2 (IL2), interferon,Granulocyte Colony-Stimulating Factor(G-CSF),Granulocyte Macrophage Colony-stimulating Factor (GM-CSF), etc.
10. Use of immune suppressive drugs.
11. Subject is currently taking any of the following drugs: midazolam, triazolam, terfenadine, astemizole, cisapride, pimozide, propafenone, flecainide, certain ergot derivatives (ergotamine, dihydroergotamine, ergonovine, and methylergonovine), rifampin, lovastatin, simvastatin, St. John's Wort, doxorubicin, ribavirin, coumadin.
12. Subject has significant history of cardiac, renal, neurologic, psychiatric, oncologic, endocrinologic (including diabetes mellitus), metabolic, or hepatic disease that would, in the opinion of the investigator, adversely affect his/her participation in this study.
13. Unable or unwillingness to discontinue use of specific medications implicated in drug interactions while on Lopinavir/ritonavir
14. Known hypersensitivity, allergic reactions, or intolerance to Lopinavir/ritonavir or to ritonavir in the past
15. Have previously received Lopinavir/ritonavir for more than 3 months in the past
16. Active substance or alcohol abuse, in the opinion of the principal investigator would interfere with protocol adherence
17. Unwillingness to use effective barrier contraception.
18. Experimental vaccines, to include HIV vaccines.
19. Patient who is currently enrolled in an experimental protocol, or is receiving an experimental medication.
20. Patients on 2 nucleoside reverse transcriptase inhibitors(NRTIs) with an Non-nucleoside-reverse transcriptase inhibitor(NNRTI) and a protease inhibitor (PI) combination will not be allowed in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Davis, MD, Principal Investigator — University of Maryland, School of Medicine, Department of Infectious Disease
Locations (1):
- University of Maryland, Institute of Human Virology, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study received IRb approval on 12/7/05. Recruitment was difficult and the inclusion criteria was amended in November 2007 to help increase enrollment.
Groups:
- Kaletra: Lopinavir/Ritonavir (Kaletra) 400/100 mg by mouth twice a day for 48 weeks.
Period: Overall Study
Arm/Group | Kaletra
Started | 3
Completed | 2 (One subject was withdrawn at month 9 because he was considered an immunologic failure on study.)
Not Completed | 1
Not completed — immunologic failure | 1

BASELINE CHARACTERISTICS:
Groups:
- Kaletra: Lopinavir/Ritonavir (Kaletra) 400/100 mgby mouth twice a day for 48 weeks
Arm/Group | Kaletra
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in CD4 Cell Count From Baseline, and at 6 and 12 Months
Time Frame: 6 and 12 months
Population: 3 patients enrolled but study terminated early due to lack of enrollment at other sites, thus unable to carry out full data analysis.Unable to report any data because original PI retired and have no access to records.
Arm/Group | Kaletra
Number analyzed (Participants) | 0

2. Primary Outcome: Changes From Baseline in CD4 Cell Percentage at 6 and 12 Months
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 1
Groups:
- Kaletra: lopinavir/ritonavir 400/100mg tablets by mouth twice a day for 48 weeks
Arm/Group | Kaletra
Number analyzed (Participants) | 0

3. Primary Outcome: Changes From Baseline in CD4 Cell Count at 6 and 12 Months
Description: Baseline Will be Defined as the Mean of 2 Values Obtained Prior to the Medication Switch (for Analysis Purposes, the CD4 Cell Counts at 6 and 12 Months Will be Defined by the Mean of the CD4 Cell Counts Obtained at Months 3, 6 or 9, 12, Respectively).
Time Frame: 6 and 12 months
Population: as for outcome 1
Arm/Group | Kaletra
Number analyzed (Participants) | 0

4. Primary Outcome: Changes in Slope of CD4
Description: Changes in Slope of CD4 as Assessed 6 Months Prior to the Lopinavir/Ritonavir Switch (baseline). Compared to 6-12 Month Intervals Post Initiation of Lopinavir/Ritonavir (Slope 1-6 Months, 1-12 Months)
Time Frame: 6 and 12 months
Population: as for outcome 1
Arm/Group | Kaletra
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse Event Reporting will be collected at each study visit.
Arm/Group | Kaletra
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
We screened and enrolled a total of three participants. Two of the three participants completed the study. Unable to meet the stated goals of the study, it was decided that it should be closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes